CLINICAL TRIAL: NCT07109323
Title: Clinical Study on the Safety and Efficacy of Autologous Hematopoietic Stem Cell Transplantation Combined With BCMA-CAR-T in the Treatment of Ultra-high Risk Multiple Myeloma
Brief Title: Autologous Transplantation Combined With BCMA CAR-T in the Treatment of UHR-MM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025026
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Ultra High Risk mm (uhr-mm), 18-70 Years Old, Suitable for ASCT. And Meet Any of the Following uhr-mm Definitions; Cytogenetics Ultra High Risk; Primary Refractory; Early Progression; Plasma Cell Leukemia; Non Paraosseous Extramedullary Infiltration; R2-ISS-IV /MPSS-IV
MeSH Terms: conditions — Disease Progression; Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART (Experimental): BCMA-CART was reinfused at a dose of 1.0-2.0 × 10 ^ 6 CAR-T cells/ kg on day +3 (± 1 day) after autologous hematopoietic stem cell reinfusion.
  Interventions: Drug: BCMA CART

INTERVENTIONS:
Drug: BCMA CART — Bcma-cart was reinfused at a dose of 1.0-2.0 × 10 ^ 6 / kg on day +3 (± 1 day) after autologous hematopoietic stem cell reinfusion.

SUMMARY:
To evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation (ASCT) combined with BCMA-CART in the treatment of UHR-MM.

DETAILED DESCRIPTION:
This study is a single center, prospective clinical study initiated by researchers to evaluate the safety and efficacy of autologous hematopoietic stem cell transplantation combined with BCMA CAR-T in the treatment of ultra high risk multiple myeloma (UHR-MM).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

Ultra high risk mm (UHR-MM), 18-70 years old, suitable for ASCT. And meet any of the following definitions of UHR-MM: 1) cytogenetic ultra-high risk, which meets any of the following conditions, including: del(17p)≥60%； Two or more cytogenetic features: TP53 mutation, del (17p) or p53 deletion, t (4; 14), t (14; 16), t (14; 20), 1q21 gain or amplification, 1p deletion, myc translocation (deletion or copy number abnormality: ≥ 20% is positive; translocation: ≥ 10% is positive); 2) Primary refractory (first-line induction therapy based on standard three drug combination: 2 courses < Mr, 4 courses < PR); 3) Early progression (the best first-line treatment response of the regimen based on the standard three drug combination is maintained for less than 6 months); 4) Plasma cell leukemia (meeting the diagnostic criteria of mm at the initial diagnosis, and the proportion of peripheral plasma cells ≥ 5%); 5) Non paraosseous extramedullary infiltration; 6) R2-iss-iv /mpss-iv.

1. The subjects voluntarily participated in the study and signed the informed consent form (ICF) by themselves or their legal guardians;
2. The subject must have proper organ function and meet all the following inspection results:

Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Creatinine clearance (CrCl) (Cockcroft Gault formula) ≥ 40ml/min; Prothrombin time (PT) ≤ 1.5 × ULN, partial prothrombin time (APTT) < 1.5 × ULN, international normalized ratio (INR) < 1.5 × ULN; Hemoglobin (HB) ≥ 60g/L; Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L (no growth factors such as granulocyte colony-stimulating factor [G-CSF] received within 7 days before laboratory examination in screening period); Absolute lymphocyte count (ALC) ≥ 0.5 × 10^9/L; Platelet (PLT) ≥ 50 × 10^9/L (no platelet transfusion within 7 days before laboratory examination in screening period); Left ventricular ejection fraction (LVEF) ≥ 45%; Blood oxygen saturation (SpO2) ≥ 92%; (3) The ECoG score is 0-1. See Appendix V for ECOG score; (4) Estimated survival ≥ 3 months; (5) The pregnancy test of fertile female subjects should be negative and not within the lactation period; Both female and male subjects need to take effective contraceptive tools or drugs within 24 months after cell infusion.

-

Exclusion Criteria:Subjects who have one or more of the following cannot be selected for this study:

1. Have a history of allergy to any component in cell products;
2. Serious heart disease, including but not limited to:

   Myocardial infarction, cardiac angioplasty or stent implantation within 6 months before signing ICF Unstable angina Severe arrhythmia History of severe non ischemic cardiomyopathy Congestive heart failure (New York Heart Association [nyha] class III or IV), and the NYHA score is shown in Appendix II
3. History of autologous / allogeneic hematopoietic stem cell transplantation;
4. Stroke or seizure within 6 months before signing ICF;
5. Have autoimmune disease, immune deficiency or other diseases requiring immunosuppressant treatment;
6. Within 3 years before signing the ICF, patients with malignant tumors other than multiple myeloma, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, breast ductal carcinoma in situ after radical surgery, and carcinoma in situ in other parts one year after radical surgery, and there has been no treatment and no recurrence in the screening period Signs;
7. The presence of uncontrolled active infection;
8. Unstable systemic diseases judged by the investigator: including but not limited to serious liver, kidney or metabolic diseases requiring drug treatment;
9. Any of the following conditions exist within 1 week before lymphocyte collection:

   The detection value of hepatitis B virus (HBV) DNA in peripheral blood was higher than the lower limit of detection Hepatitis C virus (HCV) antibody positive and peripheral HCV-RNA positive Human immunodeficiency virus (HIV) antibody positive Syphilis antigen or antibody positive Cmv-dna positive
10. More than 5mg/d prednisone (or equivalent amount of other corticosteroids) was applied within 1 week before lymphocyte collection Vegan);
11. Have used any car-t cell products or other genetically modified T cell therapies;
12. Received BCMA targeted therapy;
13. Have a history of live vaccination within 4 weeks before signing ICF;
14. Have a history of alcohol abuse, drug abuse or mental illness;
15. Other researchers consider it inappropriate to participate in this study. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2030-03-02 (Estimated)

PRIMARY OUTCOMES:
MRD negative rate at 3 month after treatment of ASCT+CAR-T | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No